CLINICAL TRIAL: NCT06478264
Title: Efficacy and Safety of Adebrelimab Combined With Chemoradiotherapy in the Treatment of Esophageal Small Cell Carcinoma: a Single-arm, Multicenter, Phase II Clinical Study
Brief Title: A Study of Adebrelimab Combined With Chemoradiotherapy in the Treatment of Esophageal Small Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhangzhou Municipal Hospital (Other)
Responsible Party: Principal Investigator, Weilin Chen, Head of radiation oncology, Zhangzhou Municipal Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVENT-ESCC
Record Dates: First submitted 2024-06-23; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Esophageal Small Cell Carcinoma
Keywords: Esophageal Small Cell Carcinoma; Adebrelimab; chemoradiotherapy
MeSH Terms: interventions — Etoposide; Cisplatin; Carboplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): EP regimen:Etoposide and Cisplatin or Carboplatin
  Cohort A: Stage I-IVa , EP combined with adebrelimab induction therapy for 2 cycles, sequential thoracic radiotherapy combined with EP chemotherapy for 2 cycles, and adebrelimab immunomaintenance therapy until PD or over 1 year.Thoracic radiotherapy regimen : prescription dose: PTV 50Gy/25f.
  Cohort B: Stage IVb , EP regimen combined with adebrelimab injection immunotherapy for 4 cycles, PR or SD patients evaluated for 3 months, followed by chest radiotherapy, and adebrelimab immunization continued until PD or full 1 year.Chest radiotherapy : prescribed dose: PTV 30Gy/10f.
  Interventions: Drug: Etoposide; Drug: Cisplatin; Drug: Carboplatin; Drug: Adebrelimab; Radiation: radiotherapy

INTERVENTIONS:
Drug: Etoposide — 100mg/m^2, intravenous infusion for 1-3 days,21 days/cycle, 4 cycles
Drug: Cisplatin — 25mg/m^2 ,intravenous infusion for 1-3 days ,21 days/cycle, 4 cycles
Drug: Carboplatin — Carboplatin (AUC = 5) on 1 Day,21 days/cycle, 4 cycles ;
Drug: Adebrelimab — 1200mg adebrelimab was given intravenously on 2 day after chemotherapy,21 days/cycle, continuous use.
  Other Names: SHR-1316
Radiation: radiotherapy — Stage I-IVa , prescription dose: PTV 50Gy/25f. Stage IVb ,prescribed dose: PTV 30Gy/10f.

SUMMARY:
To evaluate the efficacy and safety of adebrelimab combined with chemoradiotherapy in the treatment of esophageal small cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

* 1. Sign a written informed consent to join the study voluntarily;
* 2. Histologically or cytologically confirmed patients with small cell carcinoma of the esophagus staging T1N0M0 but unable to tolerate surgery or refusing surgery and patients staging T2-4N0-3M0 [according to AJCC 8th edition TNM criteria];
* 3. Age 18-75 years old, male or female;
* 4. ECOG PS 0-1;
* 5. No previous systemic treatment for esophageal small cell carcinoma;
* 6. At least one measurable lesion (according to RECIST1.1 criteria);
* 7. Normal functioning of major organs, including:

  1. Blood routine examination (no blood component, cell growth factor, white enhancer, platelet enhancer, anemia correction drugs are allowed within 14 days before the first use of the study drug) :

     White blood cell count ≥4.0×10^9/L

     Neutrophil count ≥1.5×10^9/L

     Platelet count ≥80×10^9/L

     Hemoglobin ≥90 g/L
  2. Blood biochemical examination:

     Total bilirubin ≤1.5×ULN

     ALT≤2.5 x ULN, AST≤2.5 x ULN,

     Serum creatinine ≤1.5×ULN, or creatinine clearance ≥50mL/min (Cocheroft-Gault formula, see Annex 2)
  3. Coagulation function:

International Standardized ratio (INR) ≤1.5×ULN

Activated partial thromboplastin time (APTT) ≤1.5×ULN

* 8. Patients must submit pre-treatment tumor tissue samples during the study period;
* 9. Expected survival ≥12 weeks;
* 10. Fertile female subjects are required to take a serum or urine pregnancy test with a negative result within 72 hours before starting the study drug administration, and to use effective contraception (such as an IUD, contraceptive pill or condom) during the trial period and for at least 3 months after the last drug administration; For male subjects whose partners are women of reproductive age, effective contraception should be used during the trial period and within 3 months after the last dose;
* 11. The subjects had good compliance and cooperated with follow-up visits.

Exclusion Criteria:

* 1. Esophageal perforation or hematemesis;
* 2. Uncontrolled pleural effusion, pericardial effusion or ascites requiring repeated drainage;
* 3. Uncontrolled hypercalcemia or symptomatic hypercalcemia;
* 4. Other malignancies diagnosed within 5 years prior to the first use of the investigational drug, except malignancies with a low risk of metastasis or death (5-year survival > 90%), such as adequately treated skin basal cell carcinoma or squamous cell skin cancer or cervical carcinoma in situ, may be considered for inclusion;
* 5. History of any active autoimmune disease or autoimmune disease, including but not limited to: interstitial pneumonia, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (may be considered after hormone replacement therapy); Patients with psoriasis or childhood asthma/allergies in complete remission without any intervention as adults may be considered for inclusion, but patients requiring medical intervention with bronchodilators may not be included;
* 6. Previously received immune checkpoint blocking therapy;
* 7. Subjects who required systemic corticosteroids (> 10 mg/ day effective dose of prednisone) or other immunosuppressive agents within 14 days prior to initial dosing or during the study period. However, in the absence of active autoimmune disease, subjects were allowed to use topical or inhaled steroids and adrenal hormone replacement therapy at a dose ≤10 mg/ day of prednisone effectiveness.
* 8. There are clinical symptoms or diseases of heart that are not well controlled, including but not limited to: (1) NYHA grade II or above heart failure, (2) unstable angina pectoris, (3) myocardial infarction within 1 year, (4) Clinically significant supraventricular or ventricular arrhythmias that are not well controlled without or after clinical intervention;
* 9. Poor nutritional status, BMI < 18.5 Kg/m^2; If it is corrected before enrollment after symptomatic nutritional support, it can continue to be considered for enrollment after evaluation by the principal investigator;
* 10. Adverse events greater than grade 2 caused by treatment received before the first use of the investigatory drug that have not recovered (i.e., become grade 1 or reach baseline level), and adverse events (such as neurotoxicity) that are difficult to recover quickly as determined by the investigator can be included;
* 11. History of allergy to any component of adbelimab, etoposide, cisplatin or carboplatin;
* 12. A history of immunodeficiency, including HIV testing positive, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation or allogeneic bone marrow transplantation;
* 13. Severe infections (CTCAE > Grade 2), such as severe pneumonia requiring hospitalization, bacteremia, and infection complications, occurred within 4 weeks prior to the first use of the study drug; Baseline chest imaging indicated active pulmonary inflammation, signs and symptoms of infection within 14 days prior to the first use of the study drug, or the need for oral or intravenous antibiotic treatment, except in cases of prophylactic antibiotic use;
* 14. Patients found to have active pulmonary tuberculosis infection through medical history or CT examination, or had a history of active pulmonary tuberculosis infection within 1 year before enrollment, or had a history of active pulmonary tuberculosis infection more than 1 year ago without formal treatment;
* 15. Hereditary bleeding tendency or blood clotting dysfunction. There were clinically significant bleeding symptoms or definite bleeding tendencies within 3 months prior to enrollment, such as hemorrhagic gastric ulcer, stool occult blood ++ or above at baseline;
* 16. Active hepatitis B (HBV DNA≥2000 IU/mL or 10^4 copies/mL), hepatitis C (hepatitis C antibody positive and HCV RNA higher than the lower limit of assay);
* 17. Pregnant or lactating women;
* 18. The investigator determined that there were other factors that might have led to the forced termination of the study, such as other serious medical conditions (including mental illness) requiring co-treatment, alcohol, substance abuse, family or social factors, and factors that might have affected the safety or adherence of the subjects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-13 (Estimated); Primary Completion 2026-07-13 (Estimated); Study Completion 2027-07-13 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 1 year
  Refers to the proportion of all subjects with a best overall result (BOR) of complete remission (CR) or partial remission (PR) as rated according to RECIST 1.1 criteria. If efficacy of CR or PR is achieved, subjects must be confirmed not less than 4 weeks ± 7 days after the initial evaluation.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 1 year
  Refers to the proportion of all subjects with a best overall result (BOR) of complete remission (CR), partial remission (PR), and stable disease (SD) as rated according to RECIST 1.1 criteria.
Progression-free survival (PFS) | 1 year
  PFS was defined as the date from which the subject was first given medication to the date when tumor progression (as assessed by the criteria, with or without continued treatment) was first recorded or the date of death from any cause, whichever came first.
Overall survival (OS) | 2 years
  Defined as the time between the date of first dose and the death of the subject due to all causes. Subjects who were alive at the last follow-up visit had OS counted as data censored at the time of the last follow-up visit. The OS of subjects who were lost to follow-up was counted as data censored at the time of last confirmed survival prior to the lost follow-up. OS for data censoring was defined as the time from first dose to censoring.
One-Year Overall Survival Rate | 1 year
  It refers to the probability that a patient will survive one year after receiving treatment.
Two-Years Overall Survival Rate | 2 years
  It refers to the probability that a patient will survive two years after receiving treatment.
AE | 1 year
  Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event (AE) can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

OTHER OUTCOMES:
Explore potential biomarkers in tumor tissue | 1 year
  ORR corresponding to PD-L1 negative expression, positive expression (TPS≥1%), low expression (<10%), high expression (TPS>50%)
Explore potential biomarkers in the Peripheral Blood of Cancer Patients | 1 year
  ORR corresponding to the absolute lymphocyte count and specific T lymphocyte count in the peripheral blood of patients, as well as the composition of oxidized lipid species.

CONTACTS AND LOCATIONS:
Overall Officials: Weilin Chen, Principal Investigator — Zhangzhou Municipal Hospital; Yiming Li, Principal Investigator — First Affiliated Hospital of Xiamen University; Chong Deng, Principal Investigator — First Affiliated Hospital of Xiamen University; Shouguo Li, Principal Investigator — Zhongshan Hospital Affiliated to Xiamen University; Yuyi Lin, Principal Investigator — Xiamen Second Hospital; Qunrong Cai, Principal Investigator — The Second Affiliated Hospital of Fujian Medical University; Wenjie Cai, Principal Investigator — Quanzhou First Hospital

REFERENCES:
- [Result] Wen J, Fang S, Hu Y, Xi M, Weng Z, Pan C, Luo K, Ling Y, Lai R, Xie X, Lin X, Lin T, Chen J, Liu Q, Fu J, Yang H. Impacts of neoadjuvant chemoradiotherapy on the immune landscape of esophageal squamous cell carcinoma. EBioMedicine. 2022 Dec;86:104371. doi: 10.1016/j.ebiom.2022.104371. Epub 2022 Nov 23. PMID 36434949